CLINICAL TRIAL: NCT03509012
Title: A Phase I Multicenter Study of Immunotherapy in Combination With Chemoradiation in Patients With Advanced Solid Tumors (CLOVER)
Brief Title: Immunotherapy in Combination With Chemoradiation in Patients With Advanced Solid Tumors
Acronym: CLOVER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D933BC00001; 2017-002242-77 (EudraCT Number)
Record Dates: First submitted 2018-03-12; First posted 2018-04-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma
Keywords: Durvalumab; Chemotherapy; Radiotherapy; HNSCC; NSCLC; SCLC; locally-advanced; limited stage; first line
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — durvalumab; tremelimumab; Cisplatin; Carboplatin; Etoposide; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- HNSCC Arm 1 (Experimental): Durvalumab + cisplatin with radiation in patients with locally advanced squamous cell carcinoma of the head and neck (HNSCC)
  Interventions: Drug: Durvalumab; Drug: Cisplatin (dose level 4); Radiation: External beam radiation (dose level 1)
- NSCLC Arm 1 (Experimental): Durvalumab + cisplatin and etoposide with radiation in patients with locally advanced, unresectable (Stage III) non-small-cell lung cancer (NSCLC)
  Interventions: Drug: Durvalumab; Drug: Etoposide (dose level 1); Radiation: External beam radiation (dose level 2); Drug: Cisplatin (dose level 1)
- NSCLC Arm 2 (Experimental): Durvalumab + carboplatin and paclitaxel with radiation in patients with locally advanced, unresectable (Stage III) non-small-cell lung cancer (NSCLC)
  Interventions: Drug: Durvalumab; Drug: Carboplatin (dose level 1); Drug: Paclitaxel; Radiation: External beam radiation (dose level 2)
- NSCLC Arm 3 (Experimental): Investigator's choice of carboplatin and pemetrexed OR cisplatin and pemetrexed
  Interventions: Drug: Durvalumab; Drug: Carboplatin (dose level 2); Drug: Pemetrexed; Radiation: External beam radiation (dose level 2); Drug: Cisplatin (dose level 2)
- SCLC Arm 1 (Experimental): Patients should start with cisplatin, but if cisplatin is not tolerated, they have the option to switch to carboplatin
  Interventions: Drug: Durvalumab; Drug: Cisplatin (dose level 3); Drug: Carboplatin (dose level 2); Drug: Etoposide (dose level 2); Radiation: External beam radiation (standard)
- SCLC Arm 2 (Experimental): Patients with limited-stage small-cell lung cancer (SCLC) should start with cisplatin, but if cisplatin is not tolerated, they have the option to switch to carboplatin
  Interventions: Drug: Durvalumab; Drug: Cisplatin (dose level 3); Drug: Carboplatin (dose level 2); Drug: Etoposide (dose level 2); Radiation: External beam radiation (hyperfractionated)
- SCLC Arm 3 (Experimental): Patients should start with cisplatin, but if cisplatin is not tolerated, they have the option to switch to carboplatin. Note: Arm 3 will only be opened if the regimen in SCLC Arm 1 is safe and tolerable.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Cisplatin (dose level 3); Drug: Carboplatin (dose level 2); Drug: Etoposide (dose level 2); Radiation: External beam radiation (standard)
- SCLC Arm 4 (Experimental): Patients should start with cisplatin, but if cisplatin is not tolerated, they have the option to switch to carboplatin Note: Arm 4 will only be opened if the regimen in SCLC Arm 2 is safe and tolerable.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Cisplatin (dose level 3); Drug: Carboplatin (dose level 2); Drug: Etoposide (dose level 2); Radiation: External beam radiation (hyperfractionated)

INTERVENTIONS:
Drug: Durvalumab — IV (intravenous)
  Other Names: MEDI4736
Drug: Tremelimumab — IV
  Arms: SCLC Arm 3; SCLC Arm 4
Drug: Cisplatin (dose level 4) — IV
  Arms: HNSCC Arm 1
Drug: Cisplatin (dose level 3) — IV
  Arms: SCLC Arm 1; SCLC Arm 2; SCLC Arm 3; SCLC Arm 4
Drug: Carboplatin (dose level 1) — IV
  Arms: NSCLC Arm 2
Drug: Carboplatin (dose level 2) — IV
  Arms: NSCLC Arm 3; SCLC Arm 1; SCLC Arm 2; SCLC Arm 3; SCLC Arm 4
Drug: Etoposide (dose level 1) — IV
  Arms: NSCLC Arm 1
Drug: Etoposide (dose level 2) — IV
  Arms: SCLC Arm 1; SCLC Arm 2; SCLC Arm 3; SCLC Arm 4
Drug: Paclitaxel — IV
  Arms: NSCLC Arm 2
Drug: Pemetrexed — IV
  Arms: NSCLC Arm 3
Radiation: External beam radiation (dose level 1) — radiation therapy
  Arms: HNSCC Arm 1
Radiation: External beam radiation (dose level 2) — radiation therapy
  Arms: NSCLC Arm 1; NSCLC Arm 2; NSCLC Arm 3
Radiation: External beam radiation (hyperfractionated) — radiation therapy
  Arms: SCLC Arm 2; SCLC Arm 4
Drug: Cisplatin (dose level 1) — IV
  Arms: NSCLC Arm 1
Drug: Cisplatin (dose level 2) — IV
  Arms: NSCLC Arm 3
Radiation: External beam radiation (standard) — radiation therapy
  Arms: SCLC Arm 1; SCLC Arm 3

SUMMARY:
This is an open-label, multicenter, phase I study to evaluate the safety and tolerability of durvalumab ± tremelimumab in combination with chemoradiation in patients with advanced solid tumors

DETAILED DESCRIPTION:
This study will initially treat up to approximately 300 patients with advanced solid tumors at approximately 30 sites, worldwide. The study will be composed of a dose-limiting toxicity (DLT) assessment phase (Part A) and an expansion phase (Part B).

ELIGIBILITY:
Inclusion criteria:

* World Health Organization (WHO)/ECOG performance status of 0 or 1
* Body weight >30 kg at enrollment and treatment assignment
* At least 1 measurable lesion, not previously irradiated
* No prior exposure to immune-mediated therapy (including therapeutic anticancer vaccines)
* For patients with oropharyngeal HNSCC HPV status has to be known

Exclusion criteria:

* Patients with simultaneous primary malignancies or bilateral tumors
* Active or prior documented autoimmune or inflammatory disorders
* Brain metastases or spinal cord compression
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus (HIV; positive HIV 1/2 antibodies)
* Has a paraneoplastic syndrome (PNS) of autoimmune nature
* HNSCC cohort: Head and neck cancer that does not include unresectable, locally advanced cancer of oral cavity, larynx, oropharynx or hypopharynx. HNSCC of unknown primary are also excluded
* NSCLC and SCLC cohort: Mixed SCLC and NSCLC histology
* SCLC cohort: Extensive-stage SCLC

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Dose Limiting Toxicities (DLTs) | From first dose of durvalumab until 28 days after completion of radiation therapy
Number of subjects with Adverse Events (AEs) | From first dose of durvalumab up to 90 days after the last dose of study treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From first dose until the date of objective disease progression or death, in the absence of progression at 12, 18 and 24 months, up to 4 years.
Overall Survival (OS) | From first dose until death due to any cause through study completion, up to 4 years
Objective response rate (ORR) | From first dose until disease progression, or the last evaluable assessment in the absence of progression, assessed up to 4 years.
  Number (%) of patients with an overall response of complete response (CR) or partial response (PR).
Best objective response (BoR) | From first dose until disease progression, or the last evaluable assessment in the absence of progression, assessed up to 4 years.
  The best response based on the overall visit responses from each RECIST 1.1 assessment or the last evaluable assessment in the absence of RECIST 1.1 progression.
Duration of response (DoR) | From first dose until disease progression, or death, in the absence of progression, assessed up to 4 years.
  Time from the date of first documented response until the first date of documented progression or death in the absence of disease progression.
Disease control rate (DCR) | From first dose until disease progression, at 18 weeks and 48 weeks.
Disease-free survival (DFS) | From first dose until disease progression or death, in the absence of progression at 12, 18 and 24 months, assessed up to 4 years.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (3):
  - Research Site, Tucson, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, Houston, Texas
- Japan (2):
  - Research Site, Kōtoku
  - Research Site, Sunto-gun
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Badalona
  - Research Site, Madrid
  - Research Site, Málaga
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home